CLINICAL TRIAL: NCT01249378
Title: Metabolic Impact of the Digestion of Fat in Emulsified vs Non-emulsified Form in Lean or Obese Volunteers
Brief Title: Metabolic Impact of Fat Digestion
Acronym: LIPINFLOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Pr. Martine Laville PhD, MD, Hospices Civils de Lyon, Centre de Recherche en Nutrition Humaine -Rhône-Alpes,
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2009.563/16
Record Dates: First submitted 2010-07-13; First posted 2010-11-29 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-11

CONDITIONS: Obesity
Keywords: Nutrition; Lipid; Digestion; Endotoxemia; Inflammation; Metabolism; Stable Isotope; Obesity
MeSH Terms: conditions — Obesity; Endotoxemia; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 10 g non emulsified of milk fat (Active Comparator): They are compared using the repeated measurements taken within subjects
  Interventions: Other: All subjects receive three sequences of a standard breakfast
- 40 g non emulsified of milk fat (Active Comparator): The subjects receive three sequences of different breakfasts. They are compared using the repeated measurements taken within subjects.
  Interventions: Other: All subjects receive three sequences of a standard breakfast
- 40 g finely emulsified of milk fat (Active Comparator): The subjects receive three sequences of different breakfasts. They are compared using the repeated measurements taken within subjects.
  Interventions: Other: All subjects receive three sequences of a standard breakfast

INTERVENTIONS:
Other: All subjects receive three sequences of a standard breakfast — All subjects receive three sequences of a standard breakfast containing :
  * 10 g non emulsified
  * or 40 g non emulsified
  * or 40 g finely emulsified of milk fat with stable isotope (13C triglyceride). The administration order is determined by randomized allocation. The wash-out period is three weeks. There are not diet or exercise interventions. Only, one week before and three days after, the subjects consume neither naturally enriched in 13C foods or pre/probiotics. In addition, three days before and three days after each test, the subjects receive dietary instructions

SUMMARY:
In this study, the investigators are interested in investigating how the emulsification state and amount of fat in a meal can modify the kinetics of postprandial lipemia and inflammatory outcomes (including endotoxemia) in obese vs lean subjects.

10 lean and 10 obese volunteers will come 3 times (>3 weeks apart) at the investigation center to receive a standard breakfast containing milk fat (10 g non emulsified, or 40 g non emulsified, or 40 g finely emulsified). 13C triglyceride stable isotopes will allow to follow the metabolic fate of fatty acids and calculate lipid oxidation by breath test. Blood sampling throughout digestion will allow to measure metabolic, lipid and inflammation parameters. Stool will be analysed to determine lipid losses in faeces and to phenotype microbiota.

ELIGIBILITY:
Inclusion Criteria:

* No smokers
* BMI 18 to 35 kg/m2
* Moderate physical activity
* Safety subject during medical consultation

Exclusion Criteria:

* Medical history which may affect lipid metabolism and gut microflora (renal -cardiovascular -hepatic- endocrine-inflammatory diseases)
* Drug use that could affect lipid metabolism and gut microflora (steroids, antilipemic agent, anorectic, antibiotic)
* Inflammatory or infectious disease in the last three month
* C Reactive Protein > 20
* Prebiotic or probiotic high consumers (several times a day)
* Eating disorder
* Claustrophobic subjects

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Time of appearance of plasma triglyceride peak after ingestion of emulsified vs unemulsified fat during breakfast | four hours

SECONDARY OUTCOMES:
Kinectics of: Lipid oxidation plasma metabolite concentrations Endotoxemia and plasma markers of inflammation 13 C-fatty acid appearance in plasma | one day
  Subgroups analysis on subjects BMI amount of ingested fat and emulsified or unemulsified state of ingested fat

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon,Centre de Recherche en Nutrition Humaine Rhône-Alpes (CRNH-RA), Lyon, 165 Chemin Du Grand Revoyet, France

REFERENCES:
- [Derived] Vors C, Drai J, Pineau G, Laville M, Vidal H, Laugerette F, Michalski MC. Emulsifying dietary fat modulates postprandial endotoxemia associated with chylomicronemia in obese men: a pilot randomized crossover study. Lipids Health Dis. 2017 May 25;16(1):97. doi: 10.1186/s12944-017-0486-6. PMID 28545546
- [Derived] Vors C, Pineau G, Drai J, Meugnier E, Pesenti S, Laville M, Laugerette F, Malpuech-Brugere C, Vidal H, Michalski MC. Postprandial Endotoxemia Linked With Chylomicrons and Lipopolysaccharides Handling in Obese Versus Lean Men: A Lipid Dose-Effect Trial. J Clin Endocrinol Metab. 2015 Sep;100(9):3427-35. doi: 10.1210/JC.2015-2518. Epub 2015 Jul 7. PMID 26151336
- [Derived] Vors C, Drai J, Gabert L, Pineau G, Laville M, Vidal H, Guichard E, Michalski MC, Feron G. Salivary composition in obese vs normal-weight subjects: towards a role in postprandial lipid metabolism? Int J Obes (Lond). 2015 Sep;39(9):1425-8. doi: 10.1038/ijo.2015.71. Epub 2015 Apr 28. PMID 25916910
- [Derived] Vors C, Pineau G, Gabert L, Drai J, Louche-Pelissier C, Defoort C, Lairon D, Desage M, Danthine S, Lambert-Porcheron S, Vidal H, Laville M, Michalski MC. Modulating absorption and postprandial handling of dietary fatty acids by structuring fat in the meal: a randomized crossover clinical trial. Am J Clin Nutr. 2013 Jan;97(1):23-36. doi: 10.3945/ajcn.112.043976. Epub 2012 Dec 12. PMID 23235199
- See also: Related Info — http://www.crnh-rhone-alpes.fr